CLINICAL TRIAL: NCT04309409
Title: Adjuvant Nivolumab Treatment in Stage II High-risk Melanoma - A Randomized, Controlled, Phase III Trial With Biomarker-based Risk Stratification
Brief Title: Adjuvant Nivolumab Treatment in Stage II (IIA, IIB, IIC) High-risk Melanoma
Acronym: NivoMela
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Dirk Schadendorf, Director of the Department of Dermatology and the West German Tumour Centre at the University Hospital, University Hospital, Essen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-7DL
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Malignant Melanoma Stage II
Keywords: Stage II malignant melanoma; patients having undergone surgery; IIA melanoma; IIB melanoma; IIC melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Patients with a risk score of > 0.0 (HR 1.48, 1.11-1.98) corresponding to high risk of relapse will be randomized at a ratio of 2:1 to receive either nivolumab as adjuvant treatment (arm A) or observation only (arm B).
  All screened patients with a risk score of ≤ 0.0 who are not eligible for randomization will be followed for RFS, DMFS and OS for at least 5 years according to German Follow-up guidelines (Arm C).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nivolumab (Arm A) (Experimental): Patients with a risk score of > 0.0 corresponding to high risk of relapse (randomized):
  Nivolumab will be applied at a flat dose of 480 mg given as 60-minute iv infusion every 4 weeks for 12 doses over 1 year. Afterwards these patients will receive intense clinical follow up according German Follow up guidelines.
  Interventions: Drug: Nivolumab
- Observation, High Risk (Arm B) (No Intervention): Patients with a risk score of > 0.0 corresponding to high risk of relapse (randomized):
  Control group (observation only). These patients will receive intense clinical follow up but no further specific therapy according German Follow up guidelines.
- Observation, Low Risk (Arm C) (No Intervention): Patients with a risk score of ≤ 0.0 corresponding to low risk of relapse who are not eligible for randomization:
  These patients will receive intense clinical follow up but no further specific therapy according German Follow up guidelines. Documentation of clinical outcome of these patients.

INTERVENTIONS:
Drug: Nivolumab — 480 mg nivolumab fixed dose given as 60-minute iv infusion every 4 weeks for 12 doses over 1 year
  Other Names: Opdivo
  Arms: Nivolumab (Arm A)

SUMMARY:
Stage II patients with primary surgical treatment of cuMM are often at risk for recurrence of their disease. This risk may be reduced by adjuvant systemic treatment. Due to toxicities of adjuvant therapies the aim is to identify patients at high risk for relapse and to administer adjuvant treatment only to these patients. Thus an optimal balance between insufficient treatment vs. overtreatment has to be found.

To define these patients a prognostic biomarker test will be used in addition to conventional AJCC staging. AJCC staging takes into account several prognostic factors. However, to subdivide stage II melanoma patients into having a low or high risk for relapse further methods are needed.

This clinical trial will evaluate whether adjuvant nivolumab treatment will improve relapse-free survival (RFS) in patients with stage II high-risk melanoma as compared to observation only. The randomized approach of this trial offers the most objective method with the least influence of bias. Since patients with stage II melanoma are usually not receiving adjuvant treatment, no patient will be undertreated in case of randomization into observational arm.

DETAILED DESCRIPTION:
The NivoMela trial is a randomized, controlled, prospective, multi-center national phase III trial with biomarker-based risk stratification.

Stage II melanoma patients having undergone surgery of the malignant melanoma will be screened using the MelaGenix GEP score to identify patients at high risk for relapse. It is expected, that 61% of screened patients will belong to this group.

Patients with a risk score of > 0.0 (HR 1.48, 1.11-1.98) corresponding to high risk of relapse will be randomized at a ratio of 2:1 to receive either nivolumab as adjuvant treatment (arm A) or observation only (arm B).

Stratification factors for randomization are:

1. Tumor stage: IIA versus IIB versus IIC
2. Gender: Female versus Male
3. Site of primary tumor: extremities versus trunk versus head &neck

All screened patients with a risk score of ≤ 0.0 who are not eligible for randomization will be followed for RFS, DMFS and OS for at least 5 years according to German Follow-up guidelines (Arm C).

Various factors that could potentially predict clinical response and incidence of AEs to treatment with nivolumab will be investigated in peripheral blood and tumor specimen taken at baseline. Data from these investigations will be evaluated for associations with clinical efficacy (eg, ORR, PFS, OS) and safety/toxicity (AE). The samples may also be used for exploratory analyses to assess biomarkers associated with melanoma and/or with immunotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of stage II (AJCCv8) melanoma arising from a primary cutaneous site after surgery therapy
2. Sentinel node biopsy (SNB) without detection of melanoma deposits
3. Randomization not later than 12 weeks after SNB procedure
4. Tumor tissue from primary tumor must be provided for biomarker analyses. In order to be randomized, a subject must be classified by MelaGenix risk analysis.
5. Men and women at the age of 18 to 80 years
6. Signed written, informed consent
7. Patients must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study
8. Minimum life expectancy of five years excluding their melanoma diagnosis
9. ECOG performance status of 0-1
10. Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to randomization:

    * White blood cells (WBC) ≥ 2000/μL
    * Neutrophils ≥ 1500/μL
    * Platelets ≥ 100 x103/μL
    * Hemoglobin ≥ 9.0 g/dL
    * Serum creatinine ≤ 1.5xUL
    * Creatinine clearance (CrCl) ≥ 40mL/min (using the Cockcroft-Gault formula)
    * AST / ALT ≤ 3 x ULN
    * Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who may have total bilirubin < 3.0 mg/dL)
11. Negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) for women of childbearing potential (WOCBP) within 72 hours prior to registration.

    Women will be considered to be of childbearing potential unless surgically sterilized (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy), or being post-menopausal for at least 24 months or being amenorrheic for > 12 months and follicle-stimulating hormone (FSH) levels ≥ 40 IU/L.
12. WOCBP and male patients with partners of childbearing potential must agree to always use a highly effective form of contraception according to CTFG during the course of this study and for at least 5 months after last dose of study medication (in Arm A only).

Exclusion Criteria:

1. History of primary uveal or mucosal melanoma
2. No access to sufficient tumor tissue of primary tumor
3. SNB procedure > 12 weeks before randomization
4. Prior active malignancy within the previous 3 years except for locally curable cancers that have been apparently cured, such as: basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the prostate, cervix, or breast. Exception: Participants with a history of non-ulcerated cutaneous/acral primary melanoma <1 mm in depth with no nodal involvement are allowed in this trial.
5. Prior or planned therapy with Interferon alpha, CTLA4 or PD-1 / PD L1 antibodies
6. Use of any investigational or non-registered product (drug or vaccine) other than the study treatment
7. Administration of live vaccines within 4 weeks before start of study therapy
8. Any immunosuppressive therapy given within the past 30 days
9. Active psychiatric or addictive disorders that may compromise his/her ability to give informed consent or to comply with the trial procedures
10. Active immune deficiencies or significant autoimmune disease
11. Serious cardiac, gastrointestinal, hepatic or pulmonary disease which would reduce life expectancy to less than five years
12. Serious intercurrent illness, requiring hospitalization
13. Other serious illnesses, e.g., serious infections requiring antibiotics or bleeding disorders
14. The patient is known to be positive for Human Immunodeficiency Virus (HIV) or other active chronic infections (HBV, HCV) or has another confirmed or suspected immunosuppressive or immunodeficient condition
15. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
16. Hypersensitivity to the active substance or to any of the excipients
17. Participation in another clinical study within the 30 days before registration
18. For female patients: Pregnancy or breast-feeding
19. For WOCBP and male patients with partners of childbearing potential: Refusal or inability to use effective means of contraception
20. Lack of availability for clinical follow-up assessments
21. Legal incapacity or limited legal capacity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Relapse-Free Survival (RFS) rates | 5 years
  Determination of efficacy of nivolumab in a biomarker-selected high-risk-enriched stage II melanoma patient population in comparison to control receiving observation only in a 2 (Arm A=nivolumab) : 1 (Arm B=observation) randomization, as measured by Relapse-Free Survival (RFS) rates at 36 and 60 months.
  RFS is defined as the time from date of registration until documented tumor progression date or date of death of any cause, whichever occurs first in all patients tested with the MelaGenix gene expression profiling (GEP).

SECONDARY OUTCOMES:
Distant metastasis-free survival (DMFS) rates | 5 years
  DMFS rates at 36 and 60 months
Melanoma-specific survival (MSS) rates | 5 years
  MSS rates at 36 and 60 months
Overall survival (OS) rates | 5 years
  OS rates at 36 and 60 months
Adverse events ≥ Grade 3 according to CTCAE Version 5.0 criteria (Safety / Toxicity) | Arm A: Until 100 days after discontinuation of dosing of the investigational product; Arm B: Until 1 year after patient´s written consent
  All adverse events ≥ Grade 3 according to CTCAE Version 5.0 criteria, that are definitely, probably, or possibly related to the administration of the investigational agent
Clinical utility/decision impact of the MelaGenix Gene Expression Profiling (GEP) Score in stratifying patients for adjuvant therapy | 5 years
  Patients with a risk score of > 0.0 (HR 1.48, 1.11-1.98) will be classified as high risk for relapse. It is expected, that 61% of screened patients will belong to this group.
  Patients with a risk score of score of ≤ 0.0 will be classified as low risk for relapse.

OTHER OUTCOMES:
Treatment-free interval (TFI) | 5 years
  Treatment-free interval (TFI) defined as the time from registration/randomization to the start of subsequent systemic therapy or the last known date alive (for those who never received subsequent cancer therapy).
Tumor mutational burden (TMB) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Schadendorf, Prof. Dr., Principal Investigator — University Hospital, Essen
Locations (20):
- Germany (20):
  - Universitätsklinikum Würzburg - Klinik für Dermatologie, Venerologie und Allergologie, Würzburg, Bavaria
  - Universitätsmedizin Rostock -Klinik und Poliklinik für Dermatologie und Venerologie, Rostock, Mecklenburg-Vorpommern
  - Universitätsklinikum Augsburg, Campus Süd, Augsburg
  - St. Josef-Hospital - Dermatologische Studienambulanz, Bochum
  - Klinikum Dortmund gGmbH - Dermatologie, Dortmund
  - Universitätsklinik Carl Gustav Carus der Technischen Universität Dresden - Klinik und Poliklinik für Dermatologie, Dresden
  - HELIOS Klinikum Erfurt, Erfurt
  - University Hospital Essen, Department of Dermatology, Skin Cancer Center, Essen
  - Universitätsklinikum Freiburg - Klinik für Dermatologie und Venerologie, Freiburg im Breisgau
  - Universitätsklinikum Gießen und Marburg GmbH - Klinik für Dermatologie und Allergologie, Giessen
  - Universitätsklinikum Hamburg-Eppendorf - Hauttumorzentrum, Hamburg
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel - Dermatologie, Kiel
  - Universitätsklinikum Leipzig - Klinik u. Poliklinik f. Dermatologie, Venerologie u. Allergologie, Leipzig
  - Universitätsklinikum Mannheim - Klinik f. Dermatologie, Venerologie u. Allergologie, Mannheim
  - Klinikum der Universität München - Klinik und Poliklinik für Dermatologie und Allergologie, München
  - Universitätsklinikum Münster - Zentrale Studienkoordination für innovative Dermatologie (ZID), Münster
  - Fachklinik Hornheide - Internistische Onkologie, Münster
  - Klinikum Nürnberg Nord - Hautklinik, Nuremberg
  - Harzklinikum Dorothea Christiane Erxleben - Klinik für Dermatologie & Allergologie, Quedlinburg
  - Universitätsklinikum Tübingen - Dermatoonkologie, Tübingen

IPD SHARING:
Plan to Share IPD: No